CLINICAL TRIAL: NCT07217587
Title: Efficacy and Safety of Nipocalimab vs Efgartigimod for Patients With Generalized Myasthenia Gravis in a Randomized, Open-label, Phase 3b, Interventional Trial Including Within Class Switching From Efgartigimod to Nipocalimab
Brief Title: Comparative Efficacy of Nipocalimab and Efgartigimod in Participants With Generalized Myasthenia Gravis
Acronym: EPIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80202135MYG3002; 80202135MYG3002 (Other: Janssen Research & Development, LLC); 2025-521130-28-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-10-15; First posted 2025-10-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1: Nipocalimab (Experimental): Participants will receive nipocalimab intravenously (IV), at a loading dose on Day 1 followed by maintenance dosing once every 2 weeks (q2w) until Week 12.
  Interventions: Drug: Nipocalimab
- Arm 2: Efgartigimod (Active Comparator): Participants will receive efgartigimod IV, once a week for 4 weeks starting from Day 1. Eligible participants will be given the option to switch to Arm 3 between Week 4 and Week 12.
  Interventions: Drug: Efgartigimod
- Arm 3: Treatment Switch (Nipocalimab) (Experimental): Participants previously treated with efgartigimod, who are directly enrolled in this arm, and eligible participants switching from Arm 2 will receive nipocalimab IV at a loading dose on Switch Day 1 followed by maintenance dosing q2w until Switch Week 12.
  Interventions: Drug: Nipocalimab

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered intravenously.
  Other Names: JNJ-80202135; JNJ-86507083
  Arms: Arm 1: Nipocalimab; Arm 3: Treatment Switch (Nipocalimab)
Drug: Efgartigimod — Efgartigimod will be administered intravenously.
  Arms: Arm 2: Efgartigimod

SUMMARY:
The purpose of this study is to assess how well nipocalimab works when compared to efgartigimod in participants with generalized myasthenia gravis (a condition in which body's immune system mistakenly attacks and damages the connection between nerves and muscles causing muscle weakness).

ELIGIBILITY:
Inclusion criteria:

For all arms:

* Medically stable on the basis of physical examination, medical history, vital signs, clinical laboratory tests, and 12-lead electrocardiogram (ECG) performed at screening
* Diagnosis of myasthenia gravis (MG) with generalized muscle weakness meeting the clinical criteria for generalized MG (gMG) as defined by the Myasthenia gravis foundation of America (MGFA) clinical classification class II a/b, III a/b, or IV a/b at screening and positive for acetylcholine receptor (AChR) antibodies
* Myasthenia Gravis-Activities of Daily Living (MG-ADL) score of greater than or equal to (>=) 5 with less than (<) 50% of symptoms coming from ocular MG-ADL sub-scores at study screening and baseline (Day 1) visits

Criteria specific to Arms 1 and 2 only:

- Has suboptimal response to current stable therapy for gMG according to the investigator or has discontinued corticosteroids and/or immunosuppressants/immunomodulators including eculizumab or other novel approved immune agents at least 4 weeks prior to baseline due to intolerance or lack of efficacy

Criteria specific to Arm 3:

- Treatment with efgartigimod IV or subcutaneous (SC) for >=1 cycle, and the final cycle is consistent with product information

Exclusion criteria:

* Any confirmed or suspected clinical immunodeficiency syndrome not related to treatment of his/her gMG, or has a family history of congenital or hereditary immunodeficiency unless confirmed absent in the participant
* Had a thymectomy within 1 year prior to baseline, or thymectomy is planned during the study
* Currently has a malignancy or has a history of malignancy within 3 years before baseline

Criteria specific to Arms 1 and 2 only:

- Has received treatment for MG with an FcRn-targeting therapy

Criteria specific to Arm 3 only:

- Is currently taking IgG monoclonal antibody therapeutics, or Fc-conjugated therapeutic agents, including factor or enzyme replacement, with the exception of efgartigimod

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-09-28 (Estimated); Study Completion 2028-09-04 (Estimated)

PRIMARY OUTCOMES:
Arms 1 and 2: Averaged Mean Percent Change from Baseline in Total Immunoglobulin G (IgG) Levels Over Weeks 8, 10 and 12 | Baseline, Weeks 8, 10 and 12
  Average mean percent change from baseline in total IgG levels over Weeks 8 , 10 and 12 will be reported.

SECONDARY OUTCOMES:
Arms 1 and 2: Averaged Mean Change from Baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) Total Score Over Weeks 8, 10 and 12 | Baseline, Weeks 8, 10 and 12
  Average mean change from baseline in MG-ADL total score over Weeks 8, 10 and 12 will be reported. The MG-ADL provides a rapid assessment of the participant's MG symptom severity. Eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, eyelid droop) are rated on a 4-point scale: 0 (no impairment) to 3 (severe impairment). The total score will be sum of eight function scores and can range from 0 to 24. A higher score indicates greater symptom severity.
Arms 1 and 2: Mean Percent Change from Baseline in Total IgG Between Arm 1 at EoT and Arm 2 at EoC Based on Clinical Evaluation | Baseline, EoT (for Arm 1) and EoC (Arm 2) up to Week 12
  Mean percent change from baseline in total IgG between Arm 1 at end of treatment (EoT) and Arm 2 at end of cycle (EoC) based on clinical evaluation will be reported. EoC based on clinical evaluation is defined as the timepoint at which after completion of one cycle of efgartigimod, based on MG-ADL score clinical criteria, the treatment decision would be made to start a second cycle of efgartigimod, an MG rescue medication, or Week 12/EoT, whichever occurs first.
Arms 1 and 2: Mean Percent Change from Baseline in MG-ADL Total Score Between Arm 1 at EoT and Arm 2 at EoC Based on Clinical Evaluation | Baseline, EoT (for Arm 1) and EoC (Arm 2) up to Week 12
  Mean change from baseline in MG-ADL total score between Arm 1 at EoT and Arm 2 at EoC based on clinical evaluation will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arms 1 and 2: Mean Percent Change from Baseline in Total IgG Levels at Week 8 | Baseline and Week 8
  Mean percent change from baseline in total IgG levels at Week 8 will be reported.
Arms 1 and 2: Mean Change from Baseline in MG-ADL Total Score at Week 8 | Baseline and Week 8
  Mean change from baseline in MG-ADL total score at Week 8 will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arms 1 and 2: Averaged Mean Change from Baseline in Quantitative Myasthenia Gravis (QMG) Total Score Over Weeks 8 and 12 | Baseline, Weeks 8 and 12
  Average mean change from baseline in QMG total score over Weeks 8 and 12 will be reported. The QMG test is a standardized quantitative strength assessment comprising 13 components. The quantitative results of each strength component are mapped to the following 4-point scale: 0 = None, 1 = Mild, 2 = Moderate and 3 = Severe. The total score can range from 0 to 39. A higher score indicates greater weakness.
Arms 1 and 2: Mean Percent Change from Baseline in QMG Total Score Between Arm 1 at EoT and Arm 2 at EoC Based on Clinical Evaluation | Baseline, EoT (for Arm 1) and EoC (Arm 2) up to Week 12
  Mean change from baseline in QMG total score between Arm 1 at EoT and Arm 2 at EoC based on clinical evaluation will be reported. The QMG test is a standardized quantitative strength assessment comprising 13 components. The quantitative results of each strength component are mapped to the following 4-point scale: 0 = None, 1 = Mild, 2 = Moderate and 3 = Severe. The total score can range from 0 to 39. A higher score indicates greater weakness.
Arms 1 and 2: Mean Change from Baseline in QMG Total Score at Week 8 | Baseline and Week 8
  Mean change from baseline in QMG total score at Week 8 will be reported.
Arms 1 and 2: Percentage of Participants Maintaining >= 2-Point Improvement in MG-ADL Total Score for At Least 6 Weeks During Randomized Treatment Phase | Baseline up to Week 12
  Percentage of participants maintaining >= 2-point improvement in MG-ADL total score for at least 6 weeks during the 12 week randomized treatment phase between Arms 1 and 2 will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arms 1 and 2: Percentage of Participants Maintaining >= 2-Point Improvement in MG-ADL Total Score for At Least 8 Weeks During Randomized Treatment Phase | Baseline up to Week 12
  Percentage of participants maintaining >= 2-point improvement in MG-ADL total score for at least 8 weeks during the 12 week randomized treatment phase between Arms 1 and 2 will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arms 1 and 2: Percentage of Participants Maintaining >= 2-Point Improvement in MG-ADL Total Score for 50% of Postbaseline Observations | Baseline, Week 2 up to Week 12
  Percentage of participants maintaining >= 2-point improvement in MG-ADL total score for at least 50% of study duration between Arms 1 and 2 will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arms 1 and 2: Percentage of Participants Maintaining >= 2-Point Improvement in MG-ADL Total Score for 75% of Postbaseline Observations | Baseline, Week 2 up to Week 12
  Percentage of participants maintaining >= 2-point improvement in MG-ADL for at least 75% of study duration between Arms 1 and 2 will be reported.
Arms 1 and 2: Percentage of Participants with MG-ADL Total Score of 0 or 1 at Week 12 | Week 12
  Percentage of participants with MG-ADL total score of 0 or 1 at end of study treatment between Arms 1 and 2 will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arm 3: Mean Percent Change in Total IgG from Switch Day 1 to Switch Week 12 | Switch Day 1 to Switch Week 12
  Mean percent change in total IgG from pre-nipocalimab exposure to end of nipocalimab study treatment in Arm 3 will be reported.
Arm 3: Mean Change in MG-ADL Total Score from Switch Day 1 to Switch Week 12 | Switch Day 1 to Switch Week 12
  Mean change in MG-ADL total score from pre-nipocalimab exposure to end of nipocalimab study treatment in Arm 3 will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arm 3: Percentage of Participants with >= 2-Point Improvement in MG-ADL Total Score at Switch Week 12 | At Switch Week 12
  Percentage of participants with >= 2-point improvement in MG-ADL total score at switch week 12 in Arm 3 will be reported.
Arm 3: Percentage of Participants Maintaining >= 2-Point Improvement in MG-ADL Total Score for At Least 6 Weeks During Treatment Phase | Switch Day 1 up to Switch Week 12
  Percentage of participants maintaining >= 2-point improvement in MG-ADL total score while on nipocalimab for at least 6 weeks during treatment phase in Arm 3 will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arm 3: Percentage of Participants with MG-ADL Total Score of 0 or 1 at Switch Week 12 | At Switch Week 12
  Percentage of participants with MG-ADL total score of 0 or 1 at switch week 12 in Arm 3 will be reported. MG-ADL provides a rapid assessment of the participant's MG symptom severity. The total score can range from 0 to 24. A higher score indicates greater symptom severity.
Arms 1 and 2: Number of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Up to Week 20
  An AE is any untoward medical occurrence in a clinical study participant administered with a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important. Treatment-emergent AEs associated with a. infections that are severe or require IV anti-infective or operative/invasive intervention, b. events of hypoalbuminemia <20 g/L and c. serious and non-serious venous thromboembolism (VTE; deep vein thrombosis [DVT] and/or pulmonary embolism [PE]) will be considered AESIs.
Arm 3: Number of Participants with AEs, SAEs and AESIs | Up to Switch Week 20
  An AE is any untoward medical occurrence in a clinical study participant administered with a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important. Treatment-emergent AEs associated with a. infections that are severe or require IV anti-infective or operative/invasive intervention, b. events of hypoalbuminemia <20 g/L and c. serious and non-serious venous thromboembolism (VTE; DVT and/or PE) will be considered AESIs.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- United States (3):
  - SFM Clinical Research LLC, Boca Raton, Florida
  - HSHS St. Elizabeth's Hospital, O'Fallon, Illinois
  - Henry Ford Hospital, Detroit, Michigan
- Israel (2):
  - Rambam Medical Center, Haifa
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency